CLINICAL TRIAL: NCT07149025
Title: Intractable Singultus Pilot Study
Brief Title: OMT & Intractable Singultus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, J'Aimee Lippert, Associate Professor, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY 7900
Record Dates: First submitted 2025-08-20; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hiccup
Keywords: intractable singultus; chronic hiccup
MeSH Terms: conditions — Hiccup | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OMT (Experimental)
  Interventions: Procedure: Osteopathic Manipulative Therapy

INTERVENTIONS:
Procedure: Osteopathic Manipulative Therapy — 1 session of OMT
  Other Names: ONMM; OMM

SUMMARY:
This study plans to use the effects osteopathic manipulative medicine (OMM) techniques to aid in treatment of patients with symptoms of, somatic dysfunction related to, and/or a diagnosis of Intractable Singultus. The aim of our study is to document any changes in associated symptoms of Intractable Singultus before and after osteopathic manipulative treatment (OMT).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Living with daily episodes of hiccups that have lasted longer than 1 month

Exclusion Criteria:

* Any contraindications to OMT based on screening questionnaire or during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Number of Hiccups | Days 1-7 before OMT (baseline), and Days 1-7 following OMT

CONTACTS AND LOCATIONS:
Locations (1):
- MSU OMM Clinic, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: No